CLINICAL TRIAL: NCT04085562
Title: Effect of Amlodipine Versus Bisoprolol on Hypertensive Patients With End-stage Renal Disease on Maintenance Hemodialysis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Damanhour University (Other)
Responsible Party: Principal Investigator, Ahmed Youssef, Teaching assistant, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201243
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Hypertension, Renal
MeSH Terms: conditions — Hypertension, Renal | interventions — Bisoprolol; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amlodipine (Experimental): Hypertensive patients on dialysis receiving Amlodipine 5-10 mg tablet daily alone or as part of antihypertensive regimen.
  Interventions: Drug: Amlodipine 5-10 mg
- Bisoprolol (Experimental): Hypertensive patients on dialysis receiving Bisoprolol 5-10 mg tablet daily alone or as part of antihypertensive regimen.
  Interventions: Drug: Bisoprolol Fumarate 5-10 mg

INTERVENTIONS:
Drug: Bisoprolol Fumarate 5-10 mg — Bisoprolol as antihypertensive drug in patients on hemodialysis
  Arms: Bisoprolol
Drug: Amlodipine 5-10 mg — Amlodipine as antihypertensive drug in patients on hemodialysis
  Arms: Amlodipine

SUMMARY:
Hypertension is highly prevalent in hemodialysis (HD) patients and leads to increased morbidity and mortality due to cardiovascular disease(CVD). Left ventricular hypertrophy (LVH) is both a manifestation of hypertension caused end-organ damage and an independent risk factor for CVD. Evidence shows that Beta-blockers, especially of low dialyzability decrease risk of CVD and mortality. Calcium channel blockers (CCBs) were also shown to effectively control BP in the volume expanded state and reduce cardiovascular disease risk. Asymmetric dimethyl arginine (ADMA) is a uremic toxin that decreases NO synthesis and is correlated to LVH, carotid intimal thickness (CIT), CVD, and mortality. Amlodipine is shown in one study to significantly reduce ADMA level in HD patients. The purpose of this study is to determine the effect of calcium channel blocker Amlodipine compared to Beta-blocker Bisoprolol on regression of LVH, reduction of ADMA plasma level and on BP control among hypertensive patients on HD.

ELIGIBILITY:
Inclusion Criteria:

* On maintenance hemodialysis 3 times weekly for at least 3 months.
* Hypertensive as determined by predialytic BP > 140/ 90, post-dialytic > 130/80, home-measured BP >140/90, Office based BP >140/90 and/or on antihypertensive medication.

Exclusion Criteria:

* History of malignancy.
* History of significant valvular heart disease.
* Chronic congestive heart failure.
* History of coronary artery disease.
* Ongoing atrial fibrillation.
* Known drug abuse.
* Known contraindication to Bisoprolol or Amlodipine.
* History of MI
* History of Stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Mass Index | 6 months

SECONDARY OUTCOMES:
Change in ADMA Blood level | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Youssef, BSPharm, Principal Investigator — Alexandria University; Noha El-khodary, Phd, Study Director — Faculty of pharmacy, Damanhour University; Maged Wasfy, Phd, Study Director — Faculty of pharmacy, Damanhour University; Hesham Elghonemy, Phd, Study Director — University of Alexandria
Locations (1):
- El Mowassat University hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data underlying results.
Supporting Information: ICF
Time Frame: Starting 6 months after publication.
Access Criteria: * Controlled access to data.
  * Requests are made to the PI.
  * Requests are reviewed and answered by the PI.
  * Data will be provided through E-mail.

REFERENCES:
- [Derived] Youssef AM, Elghoneimy HA, Helmy MW, Abdelazeem AM, El-Khodary NM. Effect of amlodipine versus bisoprolol in hypertensive patients on maintenance hemodialysis: A randomized controlled trial. Medicine (Baltimore). 2021 Dec 23;100(51):e28322. doi: 10.1097/MD.0000000000028322. PMID 34941131